CLINICAL TRIAL: NCT07381010
Title: Caregivers' Transfer of Dementia Knowledge as Supported by Structured Retrieval Practice
Brief Title: Learn About Caring for a Person Living With Dementia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Christian University (Other)
Responsible Party: Principal Investigator, Uma Tauber, Professor, Texas Christian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-153b
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: dementia care; symptoms of dementia; caregiver knowledge
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with caregivers randomly assigned to either the treatment (intervention) or active control comparison.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be masked to study hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Retrieval Practice (SRP) intervention (Experimental)
  Interventions: Behavioral: Structured Retrieval Practice (SRP)
- Active Control Comparison (Active Comparator): Rereading
  Interventions: Behavioral: Standard Health Education

INTERVENTIONS:
Behavioral: Structured Retrieval Practice (SRP) — Our Structured Retrieval Practice (SRP) Caregiver Intervention is a web-based multi-media program designed to enhance dementia caregivers' goal-relevant memory, reduce caregiver stress, and reduce perceptions of symptom severity. The self-guided online intervention does not require supervision by a healthcare professional. Caregivers learn modules on dementia care and complete dynamic multiple-choice tests targeting practical knowledge supported with detailed, elaborative feedback to correct health misconceptions.
  Arms: Structured Retrieval Practice (SRP) intervention
Behavioral: Standard Health Education — Caregivers re-read modules on Alzheimer's Disease or related dementias (ADRD) in a webpage format, as would be available from online resources (e.g., National Institutes of Health) to mirror how most caregivers obtain information.
  Arms: Active Control Comparison

SUMMARY:
The goal of is project is to improve caregiver education about the behavioral and psychological symptoms (BPSD) of dementia. This intervention will incorporate principles from the science of learning for structuring retrieval practice to optimize learning and long-term retention of key health information. The processing-knowledge model for ADRD care predicts that enhancing health knowledge using structured retrieval practice will best support caregivers of people living with dementia (PLwD).

DETAILED DESCRIPTION:
This study consisted of a screener and two sessions. Participants began by answering screener questions to see if they qualified to participate in the study. In Session 1, participants completed measures of self-efficacy and dementia symptom severity at their own pace. Next, participants studied 4 categories of emotions and mood symptoms of ADRD (agitation, irritation, apathy, depression) in a webpage format, as would be available from online resources (e.g., National Institutes of Health) to mirror caregivers often obtain information. Study was self-paced and order of topics was randomized. Following study, caregivers were randomly assigned to the restudy group or the structured retrieval group. Those in the restudy group restudied the four categories in the same format as before, at their own pace. Those in the structured retrieval group took a self-paced practice test consisting of 8 multiple-choice questions for each of the 4-categories in a blocked fashion such that participants answered all 8 questions in one category, in a random order (e.g., apathy), before moving onto the next (e.g., agitation), and received detailed, corrective feedback following each answer to the multiple-choice questions. Participants either studied or practice retrieval for 3 practice blocks. The order of categories and questions was randomized for each participant during each practice block. Following practice, participants completed the 10-minute problem solving task. Participants then took a self-paced multiple-choice test consisting of all 32 multiple-choice questions (i.e., the same questions as in practice). After the test, participants completed a self-paced usability measure and provided demographic information.

Session 2 began two days later, and participants began by taking the same self-paced multiple-choice test as in Session 1. Next, they completed a vocabulary task, self-efficacy scale, dementia symptom severity scale, measure of health knowledge, information seeking, and provide demographic information. Finally, participants were thanked, debriefed, and compensated for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver for a person living with dementia
* Read and speak English
* Free from cognitive impairments that prevent consenting or completing experimental tasks

Exclusion Criteria:

* Technology issues (e.g., loss of internet connection)
* Not finishing the study
* Significant distractions
* Failing 2 or more attention or bot checks
* Response times 3+ standard deviations from the mean for time sensitive measures
* Completing session 1 in less than 1 hour

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Delayed test performance | 2 days after baseline
  Proportion correct on the final 2-day delayed test of symptoms and treatments of ADRD. The test was in multiple-choice format. Performance was explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.
Immediate test performance | Baseline
  Proportion correct on the immediate (approx. 10 min retention interval) test of symptoms and treatments of ADRD. The test was multiple-choice format. Performance was explored via percent correct on the test, magnitude of the retrieval practice effect on the test, and amount of forgetting.

SECONDARY OUTCOMES:
Caregiver Self-efficacy | pre-intervention and 2-days post baseline
  Caregiver self-efficacy for symptom management will be measured using the symptom subscale of the Family Caregiver Self-efficacy for Dementia Scale (Fortinsky, Kercher, & Burant, 2002), which includes 5 items. An example item is, "how certain are you right now that you can handle any problems your relative has, like memory loss, wandering, or behavior problems." Responses will be given using a 1 (not at all certain) to 10 (very certain) scale. We will expand this scale to include items that match with our content and our symptom presence, severity, and frequency measure. Specifically, participants will respond to 12 questions using a scale from 1 (not at all certain) to 10 (very certain). An example item is, "how certain are you right now that you can handle when your loved one living with dementia experiences false beliefs or delusions?" Caregiver self-efficacy will be measured twice applying a pre-test post-test design.
E-Health Literacy | 2 days after baseline
  The E-health Literacy Scale (eHEALS) Norman & Skinner, 2006 will be administered to assess perceived skills and comfort related to using internet resources for acquiring health knowledge. The scale includes 10 questions (e.g., I can tell high quality from low quality health resources on the internet). Questions require responding on a Likert sale ranging from 1 to 5 (1-strongly disagree, 2- disagree, 3-undecided, 4-agree, 5-strongly agree; 1-not useful at all, 2-not useful, 3-unsure, 4-useful, 5-very useful; or 1-not important at all, 2-not important, 3-unsure, 4-important, 5-very important). Composite scores will be calculated with higher scores indicate higher e-health literacy.
Letter and pattern comparison | 2 days after baseline
  Perceptual speed will be measured with the Letter Comparison Test and Pattern Comparison Test (Salthouse, 1993). The Letter Comparison Test involves 21 letter string pairs to be judged as the same or different. The Pattern Comparison Test involves 30 line patterns to be judged as the same or different. For both comparison tests, participants are given 24 seconds per test to complete as many items as possible, and performance is calculated as the number of items correct. Performance on each test will be calculated as the number of items correct, and a composite score will be calculated per participant.
Raven's Progressive Matrices | Baseline
  Non-verbal fluid intelligence will be assessed with a computerized version of Raven's progressive matrices (Raven, et al., 1998). Participants will complete 18 trials in ascending order in trial normative difficulty (Ariel, Babineau, & Tauber, 2023; adapted from Stanovich & Cunningham, 1993). For each trial, a 3 x 3 array will be displayed with 8 geometric figures. The 9th position in the bottom right-hand corner will be empty. Participants will be given 8 geometric figures from which to choose to correctly complete the array. Participants will be given 10 minutes to complete as many trials as possible. Performance will be calculated as the total number of trials correct.
Vocabulary | 2 days after baseline
  General knowledge will be assessed using a common measure of general knowledge in cognitive aging research, the Advanced Vocabulary Test I-v-4 (Ekstrom et al., 1976). Participants will be presented with a series of words and required to select the synonym for each word out of five options. Participants are given 4 min per task to complete as many words as possible (36 total problems, 8 min total). The self-paced vocabulary test is presented in a fixed order, and no feedback is provided. Performance is calculated as the number of items correct while adjusting for guessing (i.e., number of items correct - (.2 * number of items incorrect)).
Medical Health Knowledge | 2 days after Baseline
  Participants will complete the Medical Term Recognition Test (METER, Rawson et al., 2010). The METER is completed on paper. A list of 40 medical words and 40 nonwords are presented. Participants read the list of items and select the ones that they recognize as real words. Participants are instructed not to guess and to only select items they are sure were real words. Performance on the METER is calculated as the number of words correctly recognized.
Dementia Health Knowledge | 2 days after Baseline
  The Alzheimer's Disease Knowledge Scale (ADKS, Carpenter et al., 2009) will be administered, and scale composite score will be calculated. The ADKS is a 30-item true/false that has been adapted cross-culturally and used to estimate knowledge of people with varying expertise in Alzheimer's Disease. It includes 4 symptom statements (e.g., Tremor or shaking of the hands or arms is a common symptom in people with AD - False), 5 caregiving statements (e.g., People with AD do best with simple instructions giving one step at a time - True), and 4 treatment and management statements (e.g., Poor nutrition can make the symptoms of AD worse - True). Participants respond by indicating true, false, or don't know.
Performance During Learning | Baseline
  Caregivers' performance during learning will be defined as the percent correct on retrieval practice trials. Specifically, caregivers will respond to multiple choice questions during learning when engaging in retrieval practice, and learning progress will be quantified by aggregating responses across items for each block. Each multiple choice question will have 1 correct answer and 3 incorrect lures, and responses will be scored as 1 (correct) or 0 (incorrect) and then aggregated per participant. This is a quantitative measure that is standard in the science of learning and for which no validated scale is available. Performance on retrieval practice trials for the will be evaluated with item-level analysis (to explore content difficulty) and across each learning block to establish participants' rate-of-learning.
Usability Measures | Baseline
  The Perceived Usefulness (PU), Ease of Use (PEUO), Enjoyment (PNJ), Behavioral Intentions (BI), Relevance, and Output Quality (OUT) subscales of the Technology Acceptance Model (TAM) 3 scale (Venkatesh & Bala, 2008) will be administered, and scale composite score will be calculated. The subscales include 3 to 4 items. An example item from the Ease of Use scale is, "I find this system easy to use." An example item from the Enjoyment scale is, "The actual process of using the system is pleasant." Questions will be adapted for our sample. For instance, questions like, "Using the system improves my performance in my job", will be altered to read, "Using the program improves my ability to manage symptoms for an individual living with dementia." Responses to all questions will be made on a 7-point Likert scale from strongly disagree to strongly agree.
Symptom Presence, Severity, and Frequency | Pre-Intervention at Baseline and 2 days after Baseline
  The behavioral and psychological symptoms experienced by the person living with dementia will be rated by the caregiver participants using the updated version of the Neuropsychiatric Inventory Questionnaire (NPI-Q; Cummings et al., 1994; Resnick et al., 2024; Resnick et al., 2021). This measure includes 12 items that the participant will rate on presence (yes vs. no), severity (1 = mild, 2 = moderate, 3 = severe), and distress (1 = not distressing at all to 5 = extremely distressing). Perceived symptom severity will be measured twice applying a pre-test post-test design.
Demographic Characteristics | Baseline and 2 days after Baseline
  Age, gender, education level, race/ethnicity, first generation status, member of an underrepresented group, native language, socioeconomic status, occupation, zip code, relationship with individual living with Alzheimer's Disease or a related dementia (e.g., child, spouse), caregiving status and duration of caregiving, and information seeking about dementia and caregiving.
Self-reported Subjective health information | Baseline and 2 days after Baseline
  Caregivers will self-report co-morbid medical conditions for the PLwD, and will report medication use, rating of health, hospitalizations, access to health insurance for the PLwD. Caregivers will be allowed to skip any questions they desire should they prefer not to report responses to any of these questions. No measurement scale will be used for these self-report questions. Instead, these brief questions are intended to obtain general health information. Example questions include, "does the person have other chronic conditions?" "Does the person living with dementia take any prescription medications?" and "Have you gone to the hospital emergency room (ER) about the person living with dementia's health in the past year (12 months)?" Responses to these questions will be used for descriptive purposes to better understand the sample and will not be aggregated into one measure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Texas Christian University, Fort Worth, Texas
  - Virginia Wesleyan University, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code